CLINICAL TRIAL: NCT03423862
Title: Development of Predictive Biomarkers for the Rate of C-peptide Decline in Persons With Recent Onset Type 1 Diabetes
Brief Title: Development of Predictive Biomarkers
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Benaroya Research Institute (Other)
Responsible Party: Principal Investigator, Susanne Cabrera, MD, Medical College of Wisconsin
Other Study IDs: 1048169
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Type1diabetes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will be collecting stool samples as well as blood samples. Blood samples will be analyzed for HLA haplotype (a genetic sequence related to type 1 diabetes susceptibility), RNA, plasma-induced signature, simulated c-peptide by 2 hour MMTT, diabetes autoantibodies, CBC with differential, HbA1c and serum and plasma for storage. Specimens will be used and stored until none is left or until 10 years after the close of the study. Research records and data will be stored until 10 years after the close of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Mixed Meal Tolerance Test — After a 10-hour overnight fast (not eating or drinking anything except water), participants will complete a mixed meal tolerance test (MMTT):
  This involves participants drinking a "Boost" drink, like a milkshake, which will raise participants' blood sugar.
  The amount of "Boost" will be based on participants body weight, up to a maximum of 360 mL or about 1 ½ cups, and should be consumed within 5 minutes.
  An IV will be placed in participants arm and blood will be drawn from it. Blood will be drawn from the IV before and then 6 times over the next 2 hours after participants drink the "Boost".
  Other Names: MMTT

SUMMARY:
Investigators aim to further the understanding of the various factors that govern the progression of beta-cell death in individuals recently diagnosed with Type 1 diabetes (T1D). Specifically, the investigators wish to examine the utility of plasma-induced signatures and other measures as predictive biomarkers for the rate of C-peptide decline in individuals with recent onset T1D. Persistent C-peptide in individuals with T1D reflects some degree of β-cell function and is clinically associated with a reduction in both severe hypoglycemic events and microvascular complications such as diabetic nephropathy and retinopathy. There is significant heterogeneity in the rate of C-peptide decline in individuals with T1D, reflective of the complex disease process. For example, ~10% of individuals have no discernable fall in stimulated C-peptide after two years from clinical diagnosis as compared to other individuals with very rapid C-peptide decline. It is currently impossible to predict how long, and to what extent, someone will have residual C-peptide production. This complicates clinical management but also the design and interpretation of T1D β-cell preservation trials. The "gold standard" outcome measure of any T1D β-cell preservation trial is the stimulated C-peptide to a mixed meal tolerance test (MMTT). Given the variability in this measure, intervention studies must include more subjects over a longer period of time. This slows the rate of scientific discovery and increases cost. This study aims to define the governing mechanisms of post-onset T1D disease trajectory. Understanding the trajectory of the disease may lead to the development of biomarkers to predict disease progression and therapies that could reverse or prevent the development of Type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 5-17 years of age with a clinical diagnosis of T1D
2. T1D diagnosis date between 1-3 months at the time of study visit 2 (baseline visit)
3. Treatment naïve of any immunomodulatory agent
4. Receiving routine out-patient diabetes care at the CHW Diabetes Clinic

Exclusion Criteria:

1. Presence of severe, active disease that requires the use of chronic medication, with the exception of well-controlled autoimmune thyroiditis/hypothyroidism or celiac disease that is well-controlled on a gluten free diet.
2. Diabetes other than T1D
3. Chronic illness known to affect glucose metabolism
4. Psychiatric impairment, with the exception of well-controlled depression or anxiety, that will affect the ability to participate in the study
5. Female participants of child-bearing age with reproductive potential must not be knowingly pregnant
6. Any condition that, in the investigator's opinion, may compromise study participation or may confound the interpretation of the study results

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Males and females between the ages of 6 and 17 years who were diagnosed with type 1 diabetes within the 3 months prior to their first study visit, who are being treated at Children's Hospital of Wisconsin.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Predicting the honeymoon period | 3 years (the duration of the study)
  To determine if that plasma-induced transcription has utility in predicting the post-onset disease trajectory in individuals with recent onset type 1 diabetes.

SECONDARY OUTCOMES:
Establishing the relationship between baseline inflammation and other measures | 3 years (the duration of the study)
  establishing the relationship between baseline inflammation and other clinical, metabolic, genetic, hematologic, and immunologic parameters in those newly diagnosed with T1D as a means of better understanding disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Cabrera, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share samples and data with researchers at the Benaroya Research Institute, however all samples and data will be de-identified so that no PHI is shared.
Supporting Information: Study Protocol
Time Frame: 3 years (the duration of the study)
Access Criteria: Only members of the study teamwill have access to data and samples.